CLINICAL TRIAL: NCT01821339
Title: Does Residual Displacement On Standard Radiographic Views Correlate With Pelvic Ring Injury Clinical Outcome?
Brief Title: Pelvic Ring Injury
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Orthopaedic Trauma Association (Other); Prisma Health-Upstate (Other); Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00043568
Record Dates: First submitted 2013-03-27; First posted 2013-04-01 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Pelvic Ring Injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine whether displacement on one or all of the standard radiography views done within 6 months and 1 year after a pelvic injury is related to health related quality of life outcomes of patients with an isolated pelvic ring injury.

DETAILED DESCRIPTION:
This is a multicenter prospective investigation to assess the clinical outcomes of patients with an isolated pelvic ring injury. The study team plans on enrolling 60 subjects. This group will include both patients treated with and without surgical repair of the pelvic ring injury.

Concomitant injuries will be accounted in two ways first by tracking the patient's ISS (Injury Severity Score), second by tracking lower extremity fractures and lumbar spine injuries that require fixation. All patients will be enrolled within 2 weeks of injury to allow collection of outcome information asking the patients to score in a manner reflecting their perceived pre-injury level of function. The outcome instruments administered will include the short-musculoskeletal functional assessment (SMFA), the Oswestry Disability Score, Majeed Pelvis Score, and a visual analog pain score.

Patient demographics including age, income level, educational level, family support, and work status will be recorded. Additional demographic information associated with motivation of recovery from injury will be collected at the time of enrollment. Associated aspects of the injury including neurologic, urologic, or bowel injuries associated with the injury will be documented. All operative complications or wound infections involving the care of the pelvic ring injury will also be recorded. Injury classification and operative data of surgical repair will also be collected. At time of follow-up neurologic deficits, evidence of painful hardware, limb length discrepancy will be documented.

Initial radiographs and CT imaging will be taken in accordance with standard clinical care at participating centers. The decision for operative or non-operative management will be made at the discretion of the treating surgeon. At 6 months and 1 year follow-up time points, plain film radiographs including an AP Pelvis, 40 degree inlet and 40 degree outlet views will be made with a calibrated marker as described by Suzuki et al. Calibrated markers are available in standard clinical practice in Orthopaedic Surgery outpatient clinic radiology units. Use of the calibrated marker requires only that the marker, a metal ball 25mm in diameter, is included in the x-ray beam adjacent to the patient at the time of taking the radiograph. Radiographs are routine clinical practice at the follow-up time points in these patients. Outcome instruments will be administered to the patient at these time points as well.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or female age 18 year or older
2. Subject has an acute pelvic ring injury defined as sustaining fracture(s) and or dislocation(s) involving the continuity of the bony pelvic ring
3. Standard of Care CT scan and AP, Inlet, Outlet radiographs are performed done at baseline (admission)
4. Subject is willing and able to provide written informed consent for study participation with 14 days after pelvic injury
5. Subject is willing and able to comply with study protocol including return for all follow-up evaluations.

Exclusion Criteria:

1. pre-existing or injury related spinal cord injuries
2. Pre-existing arthrosis of the Sacroiliac joints or Hip joints
3. Previous pelvic ring injury
4. Type IIIB or Type IIIC open fracture other than the pelvis injury
5. no CT scan done at baseline
6. Patient does not speak or read English
7. Patient is a prisoner or is at high risk of incarceration during the follow/up period
8. Subject is likely to have problems, in the judgment of the Investigator or Research Coordinator, with maintaining follow-up (such as no fixed address, plan to move out of town in the next year, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Urgent care patients. Patients coming to the ER with a Pelvic ring Fx
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2013-03; Primary Completion 2016-02 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change in displacement on one or all of the standard radiographic views | 6 months and 1 year after injury
  Participants will be scheduled for Standard of Care follow ups at 6 months and 1 year where x-rays will be taken to assess the fracture

SECONDARY OUTCOMES:
Change in health related quality of life outcomes | Enrollment, 6 months and 1 year follow up
  Questionnaires (short-musculoskeletal functional assessment (SMFA), SF-12, the Oswestry Disability Score, Majeed Pelvis Score, and a visual analog pain score) will help the study team understand participant progress.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Olson, MD, Study Director — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States